CLINICAL TRIAL: NCT02233582
Title: Effects of Non-steroidal Anti-inflammatory Drugs (NSAIDS) on Acclimatization to High Altitude
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Ibuprofen and Altitude; IRB#14-14110 (Other: UCSF IRB)
Record Dates: First submitted 2014-09-03; First posted 2014-09-08 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: High Altitude
Keywords: altitude; mountain sickness; ibuprofen; hypoxia
MeSH Terms: conditions — Altitude Sickness; Hypoxia | interventions — Ibuprofen; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ibuprofen plus ascent to high altitude (Experimental): subjects randomized to this arm will take ibuprofen 200 mg 3 times daily during ascent and at altitude.
  Interventions: Drug: Ibuprofen
- sugar pill plus ascent to high altitude (Placebo Comparator): subjects randomized to this arm will receive the placebo
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Ibuprofen — We are simply testing if taking ibuprofen upon ascent to altitude is associated with a delayed acclimatization response to the high altitude hypoxia.
  Other Names: motrin
  Arms: ibuprofen plus ascent to high altitude
Drug: Sugar pill
  Arms: sugar pill plus ascent to high altitude

SUMMARY:
Ibuprofen is often taken by travelers to high altitude to treat the symptoms of acute mountain sickness such as headache and malaise. However, the blunting of inflammation by ibuprofen may slow the process of acclimatization to altitude, which relies on mediators of inflammation for adjustments in breathing.

The study randomizes healthy subjects to receive ibuprofen or placebo and then ascend to altitude (12,500 feet). Blood cytokines and non-invasive measurements of blood and tissue oxygen levels will be made for 48 hours at altitude. The hypothesis being tested is that subjects receiving ibuprofen will have lower blood and tissue oxygen levels after 48 hours at altitude than will placebo subjects.

DETAILED DESCRIPTION:
The study will begin with 2 days of studies in San Francisco (sea level baseline). Measurements will include non-invasive measurements of blood and tissue oxygen and venous blood draws for cytokine levels.

The altitude part of the study involves ascent to the University of California's White Mountain Research Center Barcroft Laboratory, at 12,500 feet elevation. The subjects will remain at that altitude for at least 48 hours for measurements of oxygenation and blood cytokines.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects The group of subjects in this experiment will be composed of healthy adult volunteers, over age 18 and under age 65, of any ethnic group, in good physical and mental health. We expect to enroll approximately 20 subjects. The ethnic groups represented will depend on the ethnicity of those who wish to be subjects, but no ethnic groups will be specifically sought after or rejected.

Exclusion Criteria:

Subjects will be specifically excluded according to the following criteria:

1. History of any clinically significant medical condition, particularly abnormal respiratory, cardiovascular, neurological, hematological, renal or hepatic function. A medical history and physical exam will be performed at the screening session for each subject. We will use this to determine whether the subjects are healthy and without any history of these conditions. No laboratory workup will be required
2. Regular smokers (more than 1 cigarette or cigar per day).
3. Currently active or recently treated systemic or serious local infection.
4. Recent regular use of prescription medications or regular physician care for any significant medical condition.
5. A history of high altitude pulmonary edema or high altitude cerebral edema.
6. Recent exposure to altitude (>8000 ft) in the last month or having slept at an altitude >6000 feet in the last month.
7. Inability to provide written informed consent or to be able to complete the experiment.
8. Pregnancy as determined by a urine pregnancy test if subjects believe they might be pregnant
9. Allergy to non-steroid anti-inflammatory drugs (NSAIDs) or subjects reporting history or symptoms of ulcers or other ibuprofen related contraindications discussed with the screening physician.
10. Heavy coffee drinkers or caffeine users will be advised that they may suffer rebound headache when restricted from caffeinated beverages on measurement days, and asked to carefully consider any continuing participation in the study after abstaining from caffeine during their first sea level measurements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
blood cytokine levels | on days 1 and 2 at sea level, on arrival at altitude and daily for 2 days
  venous blood sample, once a day
cerebral blood flow | once daily for 2 days at sea level, on arrival at altitude and once daily at altitude for 2 days
  optical/non-invasive measure of frontal cortex cerebral blood flow with an FDA-approved device

SECONDARY OUTCOMES:
pulse oximetry | once a day for 2 days at sea level, on arrival at altitude and daily for 2 days
  finger pulse oximetry with an FDA approved pulse oximeter

OTHER OUTCOMES:
cerebral oximetry | once daily for 2 days at sea level, on arrival at altitude and daily for 2 days
  non-invasive measurements of cerebral oxygenation with an FDA approved device
acute mountain sickness inventory | once a day at both sea level (2 days) and altitude (2 days)
  standard questionnaire concerning symptoms associated with acute mountain sickness

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, PhD/MD, Principal Investigator — University of California, San Francisco; John Feiner, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - White Mountain Research Center, Bishop, California
  - UCSF Hypoxia Research Laboratory, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared with colleagues at other University of California campuses or affiliated academic institutions. No subject identifiers will be included.
Supporting Information: Study Protocol, CSR
Time Frame: To study completion.
Access Criteria: De-identified data set only.